CLINICAL TRIAL: NCT02249416
Title: A Single Center, Open-Label, Randomised, Parallel, Multiple Dose Comparison of the Effect of Tipranavir 500 mg and Ritonavir 100 mg or Tipranavir 750 mg and Ritonavir 200 mg Twice a Day for 11.5 Days on the Pharmacokinetic Characteristics of Zidovudine 300 mg in Healthy Volunteers
Brief Title: Comparison of the Effect of Tipranavir and Ritonavir or Tipranavir and Ritonavir on the Pharmacokinetic Characteristics of Zidovudine in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1182.37
Record Dates: First submitted 2014-09-23; First posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Healthy
MeSH Terms: interventions — tipranavir; Ritonavir; Zidovudine

ARMS (2):
- TPV/RTV low + ZDV (Experimental)
  Interventions: Drug: Tipranavir (TPV) low; Drug: Ritonavir (RTV) low; Drug: Zidovudine
- TPV/RTV high + ZDV (Experimental)
  Interventions: Drug: Tipranavir (TPV) high; Drug: Ritonavir (RTV) high; Drug: Zidovudine

INTERVENTIONS:
Drug: Tipranavir (TPV) low
  Arms: TPV/RTV low + ZDV
Drug: Ritonavir (RTV) low — Norvir®
  Arms: TPV/RTV low + ZDV
Drug: Tipranavir (TPV) high — Retrovir®
  Arms: TPV/RTV high + ZDV
Drug: Ritonavir (RTV) high
  Arms: TPV/RTV high + ZDV
Drug: Zidovudine

SUMMARY:
The objective of this study was to characterize the effect of two dose combinations of tipranavir/ritonavir (TPV 500 mg/RTV 100 mg and TPV 750 mg/RTV 200 mg) administered twice daily on the pharmacokinetics (PK) of zidovudine (ZDV) and zidovudine-glucuronide (GZDV) as well as the effects of zidovudine on the pharmacokinetics of TPV/RTV

ELIGIBILITY:
Inclusion Criteria:

* Ability and willingness to give written informed consent in accordance with institutional and federal guidelines and to comply with the investigational nature of the study and the related requirements
* Healthy males or females between 18 and 60 years of age inclusive
* A Body Mass Index between 18 and 35 kg/m2
* Ability to swallow numerous large capsules without difficulty
* Reasonable probability for completion of the study, in the opinion of the investigator
* Acceptable laboratory values that indicate adequate baseline organ function are required at the time of screening. Laboratory values are considered to be acceptable if severity <= Grade 1 based on the ACTG DAIDS Grading Scale. All abnormal laboratory values > Grade 1 (e.g., CPK, amylase, triglycerides) are subject to approval by the BIPI clinical monitor
* Acceptable medical history, physical examination, ECG, and Chest X-ray are required prior to entering the study
* Willingness to abstain from alcohol for 48 hours prior to Study Day 0 and abstain from alcohol for the duration of the study. In addition, Cabernet Sauvignon must not have been ingested within 15 days prior to Day 0 (Visit 2)
* Willingness to abstain from ingesting grapefruit and grapefruit juice within 15 days of Day 0, Visit 2 and for the duration of the study
* Willingness to abstain from ingesting Seville oranges, garlic supplements, St. John's Wort, Milk Thistle, or methylxanthine-containing drinks or food (coffee, tea, cola, energy drinks, chocolate, etc.) within 72 hours of PK sampling days (Day 1 (Visit 3), Days 11-14 (Visits 5-8))
* Willingness to abstain from use of tobacco products for the duration of the study
* Urine drug screen negative for illegal non-prescription drugs
* Negative HIV serology
* Negative for Hepatitis B surface antigen and Hepatitis C

Exclusion Criteria:

* Female subjects who are of reproductive potential who:

  * Have a positive serum B-HCG at Visit 1 or 2 or,
  * Have not been using a barrier contraceptive method for at least 3 months prior to Visit 3 (Day 1) or,
  * Are not willing to use a reliable method of double-barrier contraception (such as diaphragm with spermicidal cream/jelly or condoms with spermicidal foam) during the trial and 30 days after completion / termination or,
  * Are breast-feeding
* Participation in another trial with an investigational medicine for 30 days prior to Day 0 (Visit 2)
* Ingestion of any known enzyme altering drug (such as phenothiazines, cimetidine, barbiturates, ketoconazole, fluconazole, rifampin, steroids, and herbal medications for 30 days prior to Day 0 (Visit 2)
* Ingestion of grapefruit, grapefruit juice, and Cabernet Sauvignon within 15 days prior to Day 0 (Visit 2)
* Ingestion of Seville oranges, garlic supplements, St. John's Wort, Milk Thistle, or methylxanthine-containing drinks or food (coffee, tea, cola, energy drinks, chocolate, etc.) within 72 hours of PK sampling days [Day 1 (Visit 3), Days 11-14 (Visits 5-8)]
* Ingestion of antibiotics within 10 days prior to Day 0 (Visit 2)
* Inability to comply with investigator's instructions
* History of gastrointestinal, hepatic, or renal disorders within 60 days
* History of alcohol abuse
* Current use of cigarettes defined as greater than 10 cigarettes per day
* Blood or plasma donations within 30 days prior to Day 0 (Visit 2)
* Subjects with a seated systolic blood pressure either <100 mm Hg or >150 mm Hg; resting heart rate either <50 beats/min or >90 beats/min
* Subjects with a history of any illness or allergy that, in the opinion of the investigator, might confound the results of the study or pose additional risk in administering tipranavir or ritonavir or zidovudine to the subject
* Subjects who have had an acute illness within 2 weeks prior to Day 0 (Visit 2)
* Subjects who are currently taking any over-the-counter drug within 7 days prior to Day 0, (Visit 2) or who are currently taking any prescription drug that, in the opinion of the investigator in consultation with the BIPI clinical monitor and pharmacokineticist, might interfere with either the absorption, distribution or metabolism of the test substances
* Hypersensitivity to tipranavir, ritonavir, or zidovudine

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2001-11; Primary Completion 2002-02 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma from zero time to 12 hours (AUC0-12) | Up to 12 h after drug administration
Maximum plasma concentration (Cmax) | Up to 24 h after drug administration
Drug concentration in plasma at 6 hours after drug administration (Cp6h) | Up to 6 h after drug administration
Drug concentration in plasma at 12 hours after drug administration (Cp12h) | Up to 12 h after drug administration

SECONDARY OUTCOMES:
Maximum plasma concentration at steady state (Cmax ss) | Up to 24 h after drug administration
Trough plasma concentration (Cmin) | Up to 24 h after drug administration
Mean residence time (MRT) | Up to 24 h after drug administration
Terminal half life (t1/2) | Up to 24 h after drug administration
Time of maximum concentration (tmax) | Up to 24 h after drug administration
Oral clearance (CL/F) | Up to 24 h after drug administration
Apparent volume of distribution during the terminal elimination phase (Vz/F) | Up to 24 h after drug administration
Number of participants with clinically significant changes in vital signs | Up to day 14 after first drug administration
Number of participants with abnormal findings in physical examination | Up to day 14 after first drug administration
Number of participants with abnormal changes in clinical laboratory parameters | Up to day 14 after first drug administration
Number of participants with Adverse Events | Up to day 14 after first drug administration